CLINICAL TRIAL: NCT06328790
Title: A Window Into the Mind-brain-body Interplay: Development of Diagnostic, Prognostic Biomarkers and Rehabilitation Strategies in Functional Motor Disorders
Brief Title: Study of Biomorkers and Rehabilitation Strategies in Functional Motor Disorders (FMD)
Status: Recruiting | Type: Observational
Sponsor: Michele Tinazzi, MD, PhD (Other)
Collaborators: IRCCS Ospedale San Raffaele (Other); Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Responsible Party: Sponsor-Investigator, Michele Tinazzi, MD, PhD, Principal Investigator, Universita di Verona
Organization: Universita di Verona (Other)
Other Study IDs: PNRR-MAD-2022-12376826
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Functional Motor Disorders
Keywords: Non motor symptoms; Motor symptoms; Exteroception; Interoception; Neurophysiological; MRI assessment; Diagnosis; Behavioral
MeSH Terms: conditions — Disease; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Functional Motor Disorder rehabilitation group (FMD): Patients with FMD (subject to current diagnostic criteria) will undergo experiment 3.
  Interventions: Other: Multidisciplinary Rehabilitation Training
- Healthy Controls group (HC): Healthy subjects at least 18 years old will undergo experiment 1.
  Interventions: Behavioral: Cross-sectional study on patients with FMD and healthy controls (HC)
- "Organic" Motor Disorders group: Patients with "organic" motor disorders (weakness due to peripheral neuromuscular disorders, essential tremor, or idiopathic adult-onset dystonia, all according to current diagnostic criteria) will undergo experiment 2.
  Interventions: Behavioral: Cross-sectional study on patients with FMD and patients with structural/organic diseases
- Functional Motor Disorder group (FMD): Patients with FMD (subject to current diagnostic criteria) will undergo experiment 1.
  Interventions: Behavioral: Cross-sectional study on patients with FMD and healthy controls (HC)

INTERVENTIONS:
Other: Multidisciplinary Rehabilitation Training — 34 Patients will attend the in-person 5-day rehabilitation program (2 h/day) followed by a 12-weeks telemedicine program (1 h/week).
  Other Names: Experiment 3
  Groups: Functional Motor Disorder rehabilitation group (FMD)
Behavioral: Cross-sectional study on patients with FMD and patients with structural/organic diseases — Each subject will undergo behavioural, neurophysiological, and Magnetic Resonance Imaging (MRI) tests exploring the motor, exteroceptive and interoceptive domains.
  Other Names: Experiment 2
  Groups: "Organic" Motor Disorders group
Behavioral: Cross-sectional study on patients with FMD and healthy controls (HC) — Each subject will undergo a set of behavioural, neurophysiological, and Magnetic Resonance Imaging (MRI) tests exploring the motor, exteroceptive and
  Other Names: Experiment 1
  Groups: Functional Motor Disorder group (FMD); Healthy Controls group (HC)

SUMMARY:
Functional motor disorders (FMD) are prevalent and highly disabling conditions characterized by abnormal movements (functional weakness, tremor, dystonia) significantly altered by distractive manoeuvres and incongruent with movement disorders seen in specific neurological diseases. FMDs are still misunderstood, diagnosed with delay, and not adequately treated, leading to reduced independence and high healthcare costs. Symptoms are physiologically associated with voluntary movement (distractibility, resolution with placebo) but are reported as involuntary. How this happens is yet a matter of debate. Identifying diagnostic and prognostic disease-specific biomarkers is an unmet need. The investigators will investigate motor, exteroceptive and interoceptive domains in a large cohort of FMD patients by a comprehensive set of behavioural, neurophysiological, and MRI tests. Ad-hoc eXplainable Artificial Intelligence (XAI) methods will develop disease-specific diagnostic and prognostic biomarker algorithms.

DETAILED DESCRIPTION:
Functional motor disorders (FMD) are part of the broad spectrum of functional neurological disorders characterized by abnormal movements (functional limb weakness, tremor, dystonia) significantly altered by distractive manoeuvres and incongruent with movement disorders seen in specific neurological diseases. FMDs have a high prevalence, are still misunderstood, diagnosed with a long delay, and not adequately treated, leading to high degrees of disability and poor quality of life with increasing social and economic costs. The old concept of psychological factors as the primary cause (conversion disorder) has been abandoned due to the lack of evidence about their causal role. According to a predictive coding account, the emerging idea is that symptoms and disability in FMD may depend on dysfunctions of a specific neural system integrating interoception, exteroception, and motor control. The idea underpins the investigator's proposal that FMD symptoms are perceptions of the state of the body. Besides the main pathophysiological features (abnormal attentional focus, beliefs/expectations, and sense of agency), the lived experience of symptoms and their resulting disability may depend on a specific neural system integrating motor, exteroceptive and interoceptive domains. Therefore, dysfunction within this system can cause and sustain motor and non-motor symptoms in FMD. Three-stage research will be conducted. A large cohort of patients with a definite diagnosis of FMD (n=150) and healthy controls (n=150) will be investigated by behavioural, neurophysiological, and MRI tests to collect biomarkers in the motor, exteroceptive and interoceptive domains. Computational modelling of the behavioural, neurophysiological, and MRI biomarkers will be developed through eXplainable Artificial Intelligence (XAI) methods through a data mining approach (machine learning) to implement a diagnostic algorithm biomarker (objective 1). A cohort of patients with "organic" motor disorders (n=75) will undergo the same behavioural, neurophysiological, and MRI tests belonging to the resulting biomarker-based diagnostic algorithm for validation (objective 2). Finally, the modulation of the resulting biomarker-based diagnostic algorithm after rehabilitation and the correlations of motor and non-motor symptoms (NMSs) with clinical improvement will be investigated in a sub-group of patients with FMD to explore the predictive value (objective 3). Our proposal consists of 6 work packages (WP), all integrated to deliver our stated objectives over the project's lifetime to achieve these objectives. Communication and dissemination activities will include the project's visual identity, public website, social media, videos, and press releases. Our proposal will inform the research and clinical community on disease-specific biomarkers for diagnosing and prognosis patients with FMD. The proposed approach has significant potential to disentangle some of the poorly understood features of these disorders, potentially providing a platform for more fundamental insights into brain functioning and the development of precision medicine approaches in their management. The proposed approach can also give the clinicians validated examinations to make a correct early diagnosis. This will improve the management of FMD with a positive impact on the patient's disability and the socio-economic costs of the illness.

ELIGIBILITY:
Experiments 1 and 3

Inclusion Criteria for Patients with FMD:

* Age higher or equal to 18 years
* Clinically definite diagnosis of FMD

Exclusion Criteria for Patients with FMD:

* Mini-Mental State Examination score lower or equal to 24
* Physical impairment precluding signing the informed consent for participation
* Certified other neurological and/or psychiatric comorbidities
* Contraindications for 3T MRI

Inclusion Criteria for Healthy Controls (HC)

- Age higher or equal to 18 years

Exclusion Criteria for Healthy Controls (HC) Mini-Mental State Examination score lower or equal to 24

* Physical impairment precluding signing the informed consent for participation
* Certified neurological and/or psychiatric comorbidities
* Contraindications for 3T MRI

Experiment 2

Inclusion criteria

* Age higher or equal to 18 years
* Clinically definite diagnosis of "organic" motor disorders: weakness due to peripheral neuromuscular disorders, essential tremor, or idiopathic adult-onset dystonia.
* Score>2 on the Tremor Research Group Essential Tremor Rating Assessment Scale for patients with essential tremor
* Rest tremors and other neurological signs
* Current or past exposure to tremorgenic drugs

Exclusion Criteria

* Mini-Mental State Examination score lower or equal to 24
* Physical impairment precluding signing the informed consent for participation
* Certified neurological and/or psychiatric comorbidities
* Contraindications for 3T MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experiments 1 and 3: Functional Motor Disorders Experiment 2: patients with "organic" motor disorders (weakness due to peripheral neuromuscular disorders, essential tremor, or idiopathic adult-onset dystonia)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Simplified Functional Movement Disorders Rating Scale (S-FMDRS) score | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Objective-rated validated scale to rate the duration and severity of functional motor symptoms (range: 0-54; higher = worse).
Multidimensional Fatigue Inventory Scale (MFI-20) score | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  It evaluates fatigue differentiating general, physical, reduced-activity, reduced-motivation, and mental fatigue (subscale range: 4-20; higher = worse).
Brief Pain Inventory (BPI) score | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  It evaluates pain intensity (range: 0-40; higher = worse) and interference (range: 0-70; higher = worse).
Beck Anxiety Inventory (BAI) score | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  It evaluates anxiety (range: 0-63; higher = worse).
Beck Depression Inventory (BDI-II) score | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  It evaluates depression (range: 0-63; higher = worse).
12-item Short-Form Health Survey (SF-12) score | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  The health-Related QoL will be evaluated by the Mental Health and Physical functioning of the 12-item Short-Form Health Survey (SF-12) (range: 0-100; higher = better).
Toronto Alexithymia Scale (TAS-20) score | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  It evaluates the level of alexithymia (range: 20-100; higher = worse).
Direct adn indirect index of Sensory Attenuation (SA) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Sensory attenuation (SA) will be used to collect data
Joint angle at the elbow vibrated and reproduced | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Tonic vibration reflex (TVR) will be used to collect data
N2/P2 amplitude | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Laser evoked potentials (LEP) will be used to collect data
Objective/Subjective heart rate ratio | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Heartbeat Perception Task (HPT) will be used to collect data
Cortical thickness and gray matter volumes | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Brain 3 Tesla MRI will be used to collect data
Clinical Global Impression (CGI) score | After 3 months of the intensive 5-day rehabilitation protocol (T1).
  Self-rated perception of change will be assessed with the 7-point Clinical Global Impression (CGI) scale with scores from 1 (very much improved) to 7 (very much worse).
Gait speed (cm/sec) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Gait analysis will be used to collect gait speed (cm/s).
Swing time (%) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Gait analysis will be used to collect swing time (%).
Stride time (s) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Gait analysis will be used to collect stride time (s).
Stride length (cm) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Gait analysis will be used to collect stride length (cm).
Sway area (mm2) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  An electronic monaxial stabilometric platform will be used to collect sway area (mm2).
Stance time (sec) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  An electronic monaxial stabilometric platform will be used to collect stance time (sec).
Total excursion path (mm) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  An electronic monaxial stabilometric platform will be used to collect total excursion path (mm): area of oscillations of the Center of Pressure (CoP), CoP perimeter length
Velocity of Cop displacement in the anteroposterior directions (mm/s) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  An electronic monaxial stabilometric platform will be used to collect the velocity of Cop displacement in the anteroposterior directions.
Velocity of Cop displacement in the mediolateral directions (mm/s) | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  An electronic monaxial stabilometric platform will be used to collect the velocity of Cop displacement in the mediolateral directions.
Autism spectrum Quotient (AQ) | Before the intensive 5-day rehabilitation protocol (T0)
  It is a 50-item self-report measure used to assess traits of autism in adults and adolescents aged 16 years and over (Total score: 0-50; cut-off: > 29).
Schizotypal Personality Questionnaire (SPQ) | Before the intensive 5-day rehabilitation protocol (T0)
  It is a scale for the assessment of schizotypal personality based on DSM-III-R criteria (Total score: 0-74; cut-off: < 8 & > 42).

OTHER OUTCOMES:
Number of drop-out | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  The number of dropouts before the end of treatment will be collected.
Number of patients who refuse the treatment | Before the intensive 5-day rehabilitation protocol (T0) and after 3 months of the intensive 5-day rehabilitation protocol (T1).
  Recruitment rate.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tinazzi, PhD, Principal Investigator — Universita di Verona
Locations (3):
- Italy (3):
  - Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno, Campania
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Department of Neurosciences, Biomedicine and Movement Sciences, University of Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta A, Lang AE. Psychogenic movement disorders. Curr Opin Neurol. 2009 Aug;22(4):430-6. doi: 10.1097/WCO.0b013e32832dc169. PMID 19542886
- [Background] Bhatia KP, Bain P, Bajaj N, Elble RJ, Hallett M, Louis ED, Raethjen J, Stamelou M, Testa CM, Deuschl G; Tremor Task Force of the International Parkinson and Movement Disorder Society. Consensus Statement on the classification of tremors. from the task force on tremor of the International Parkinson and Movement Disorder Society. Mov Disord. 2018 Jan;33(1):75-87. doi: 10.1002/mds.27121. Epub 2017 Nov 30. PMID 29193359
- [Background] Albanese A, Bhatia K, Bressman SB, Delong MR, Fahn S, Fung VS, Hallett M, Jankovic J, Jinnah HA, Klein C, Lang AE, Mink JW, Teller JK. Phenomenology and classification of dystonia: a consensus update. Mov Disord. 2013 Jun 15;28(7):863-73. doi: 10.1002/mds.25475. Epub 2013 May 6. PMID 23649720
- [Background] Engel AG, Myology, vol.II, 3rd ed. New York:McGraw-Hill;2004
- [Background] Piramide N, Agosta F, Sarasso E, Canu E, Volonte MA, Filippi M. Brain activity during lower limb movements in Parkinson's disease patients with and without freezing of gait. J Neurol. 2020 Apr;267(4):1116-1126. doi: 10.1007/s00415-019-09687-1. Epub 2020 Jan 2. PMID 31897599
- [Background] Cojan Y, Waber L, Carruzzo A, Vuilleumier P. Motor inhibition in hysterical conversion paralysis. Neuroimage. 2009 Sep;47(3):1026-37. doi: 10.1016/j.neuroimage.2009.05.023. Epub 2009 May 18. PMID 19450695
- [Background] Tinazzi M, Morgante F, Marcuzzo E, Erro R, Barone P, Ceravolo R, Mazzucchi S, Pilotto A, Padovani A, Romito LM, Eleopra R, Zappia M, Nicoletti A, Dallocchio C, Arbasino C, Bono F, Pascarella A, Demartini B, Gambini O, Modugno N, Olivola E, Di Stefano V, Albanese A, Ferrazzano G, Tessitore A, Zibetti M, Calandra-Buonaura G, Petracca M, Esposito M, Pisani A, Manganotti P, Stocchi F, Coletti Moja M, Antonini A, Defazio G, Geroin C. Clinical Correlates of Functional Motor Disorders: An Italian Multicenter Study. Mov Disord Clin Pract. 2020 Sep 22;7(8):920-929. doi: 10.1002/mdc3.13077. eCollection 2020 Nov. PMID 33163563
- [Background] Gandolfi M, Riello M, Bellamoli V, Bombieri F, Geroin C, Di Vico IA, Tinazzi M. Motor and non-motor outcomes after a rehabilitation program for patients with Functional Motor Disorders: A prospective, observational cohort study. NeuroRehabilitation. 2021;48(3):305-314. doi: 10.3233/NRE-201617. PMID 33780378
- [Background] Tomic A, Agosta F, Sarasso E, Petrovic I, Basaia S, Pesic D, Kostic M, Fontana A, Kostic VS, Filippi M. Are there two different forms of functional dystonia? A multimodal brain structural MRI study. Mol Psychiatry. 2020 Dec;25(12):3350-3359. doi: 10.1038/s41380-018-0222-2. Epub 2018 Aug 17. PMID 30120414
- [Background] Canu E, Agosta F, Tomic A, Sarasso E, Petrovic I, Piramide N, Svetel M, Inuggi A, D Miskovic N, Kostic VS, Filippi M. Breakdown of the affective-cognitive network in functional dystonia. Hum Brain Mapp. 2020 Aug 1;41(11):3059-3076. doi: 10.1002/hbm.24997. Epub 2020 Apr 3. PMID 32243055
- [Background] Piramide N, Sarasso E, Tomic A, Canu E, Petrovic IN, Svetel M, Basaia S, Dragasevic Miskovic N, Kostic VS, Filippi M, Agosta F. Functional MRI connectivity of the primary motor cortex in functional dystonia patients. J Neurol. 2022 Jun;269(6):2961-2971. doi: 10.1007/s00415-021-10879-x. Epub 2021 Nov 12. PMID 34773159
- [Background] Landolfi A, Ricciardi C, Donisi L, Cesarelli G, Troisi J, Vitale C, Barone P, Amboni M. Machine Learning Approaches in Parkinson's Disease. Curr Med Chem. 2021;28(32):6548-6568. doi: 10.2174/0929867328999210111211420. PMID 33430721
- [Background] Teodoro T, Koreki A, Meppelink AM, Little S, Nielsen G, Macerollo A, Ferreira JJ, Parees I, Lang A, Edwards MJ. Contingent negative variation: a biomarker of abnormal attention in functional movement disorders. Eur J Neurol. 2020 Jun;27(6):985-994. doi: 10.1111/ene.14189. Epub 2020 Apr 14. PMID 32096289
- [Background] Lorenz J, Garcia-Larrea L. Contribution of attentional and cognitive factors to laser evoked brain potentials. Neurophysiol Clin. 2003 Dec;33(6):293-301. doi: 10.1016/j.neucli.2003.10.004. PMID 14678843
- [Background] Hanzlikova Z, Kofler M, Slovak M, Vechetova G, Fecikova A, Kemlink D, Sieger T, Ruzicka E, Valls-Sole J, Edwards MJ, Serranova T. Prepulse inhibition of the blink reflex is abnormal in functional movement disorders. Mov Disord. 2019 Jul;34(7):1022-1030. doi: 10.1002/mds.27706. Epub 2019 May 2. PMID 31046188
- [Background] Gandolfi M, Fiorio M, Geroin C, Prior M, De Marchi S, Amboni M, Smania N, Tinazzi M. Motor dual task with eyes closed improves postural control in patients with functional motor disorders: A posturographic study. Gait Posture. 2021 Jul;88:286-291. doi: 10.1016/j.gaitpost.2021.06.011. Epub 2021 Jun 11. PMID 34153806
- [Background] Parees I, Brown H, Nuruki A, Adams RA, Davare M, Bhatia KP, Friston K, Edwards MJ. Loss of sensory attenuation in patients with functional (psychogenic) movement disorders. Brain. 2014 Nov;137(Pt 11):2916-21. doi: 10.1093/brain/awu237. Epub 2014 Aug 26. PMID 25161293
- [Background] Tinazzi M, Marotta A, Zenorini M, Riello M, Antonini A, Fiorio M. Movement perception of the tonic vibration reflex is abnormal in functional limb weakness. Parkinsonism Relat Disord. 2021 Jun;87:1-6. doi: 10.1016/j.parkreldis.2021.04.011. Epub 2021 Apr 20. PMID 33895678
- [Background] Grunewald RA, Yoneda Y, Shipman JM, Sagar HJ. Idiopathic focal dystonia: a disorder of muscle spindle afferent processing? Brain. 1997 Dec;120 ( Pt 12):2179-85. doi: 10.1093/brain/120.12.2179. PMID 9448573
- [Background] Fiorio M, Recchia S, Corra F, Simonetto S, Garcia-Larrea L, Tinazzi M. Enhancing non-noxious perception: behavioural and neurophysiological correlates of a placebo-like manipulation. Neuroscience. 2012 Aug 16;217:96-104. doi: 10.1016/j.neuroscience.2012.04.066. Epub 2012 May 6. PMID 22569155
- [Background] Morgante F, Matinella A, Andrenelli E, Ricciardi L, Allegra C, Terranova C, Girlanda P, Tinazzi M. Pain processing in functional and idiopathic dystonia: An exploratory study. Mov Disord. 2018 Aug;33(8):1340-1348. doi: 10.1002/mds.27402. Epub 2018 May 8. PMID 29737565
- [Background] Schandry R. Heart beat perception and emotional experience. Psychophysiology. 1981 Jul;18(4):483-8. doi: 10.1111/j.1469-8986.1981.tb02486.x. No abstract available. PMID 7267933
- [Background] Nielsen G, Ricciardi L, Demartini B, Hunter R, Joyce E, Edwards MJ. Outcomes of a 5-day physiotherapy programme for functional (psychogenic) motor disorders. J Neurol. 2015 Mar;262(3):674-81. doi: 10.1007/s00415-014-7631-1. Epub 2015 Jan 4. PMID 25557282
- [Background] Nielsen G, Buszewicz M, Stevenson F, Hunter R, Holt K, Dudziec M, Ricciardi L, Marsden J, Joyce E, Edwards MJ. Randomised feasibility study of physiotherapy for patients with functional motor symptoms. J Neurol Neurosurg Psychiatry. 2017 Jun;88(6):484-490. doi: 10.1136/jnnp-2016-314408. Epub 2016 Sep 30. PMID 27694498
- [Background] Demartini B, Bombieri F, Goeta D, Gambini O, Ricciardi L, Tinazzi M. A physical therapy programme for functional motor symptoms: A telemedicine pilot study. Parkinsonism Relat Disord. 2020 Jul;76:108-111. doi: 10.1016/j.parkreldis.2019.05.004. Epub 2019 May 3. PMID 31078400
- [Background] Guo Y, Graber A, McBurney RN, Balasubramanian R. Sample size and statistical power considerations in high-dimensionality data settings: a comparative study of classification algorithms. BMC Bioinformatics. 2010 Sep 3;11:447. doi: 10.1186/1471-2105-11-447. PMID 20815881
- [Background] Boscolo Galazzo I, Cruciani F, Brusini L, Salih A, Radeva P, Storti SF, Menegaz G. Explainable Artificial Intelligence for Magnetic Resonance Imaging Aging Brainprints: Grounds and challenges. IEEE Signal Processing Magazine, vol. 39, no. 2, pp. 99-116. 2022 March. doi: 10.1109/MSP.2021.3126573.
- [Background] Cruciani F, Brusini L, Zucchelli M, Retuci Pinheiro G, Setti F, Boscolo Galazzo I, Deriche R, Rittner L, Calabrese M, Menegaz G. Interpretable deep learning as a means for decrypting disease signature in multiple sclerosis. J Neural Eng. 2021 Jul 19;18(4). doi: 10.1088/1741-2552/ac0f4b. PMID 34181581
- [Background] Salih A, Boscolo Galazzo I, Raisi-Estabragh Z, Petersen SE, Gkontra P, Lekadir K, Menegaz G, Radeva P. A new scheme for the assessment of the robustness of Explainable Methods Applied to Brain Age estimation. IEEE 34th International Symposium on Computer-Based Medical Systems (CBMS), Aveiro, Portugal, 2021, pp. 492-497. doi: 10.1109/CBMS52027.2021.00098.
- [Background] Karch JD, Brandmaier AM, Voelkle MC. Gaussian Process Panel Modeling-Machine Learning Inspired Analysis of Longitudinal Panel Data. Front Psychol. 2020 Mar 19;11:351. doi: 10.3389/fpsyg.2020.00351. eCollection 2020. PMID 32265770
- [Derived] Gandolfi M, Sandri A, Mariotto S, Tamburin S, Paolicelli A, Fiorio M, Pedrotti G, Barone P, Pellecchia MT, Erro R, Cuoco S, Carotenuto I, Vinciguerra C, Botto A, Zenere L, Canu E, Sibilla E, Filippi M, Sarasso E, Agosta F, Tinazzi M; Group Collaborators Consortium. A window into the mind-brain-body interplay: Development of diagnostic, prognostic biomarkers, and rehabilitation strategies in functional motor disorders. PLoS One. 2024 Sep 26;19(9):e0309408. doi: 10.1371/journal.pone.0309408. eCollection 2024. PMID 39325803